CLINICAL TRIAL: NCT00512603
Title: Association Between Levels of D-Dimer, Fibrinogen and PAI-1 in Elderly Patients With Infection and Occurrence of Cardio- and Cerebro-vascular Disease After Discharge
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Asher Winder, Senior Physician, Institute of Hematology, Wolfson Medical Center, Holon, Israel. Responsible of Thrombosis & Hemostasis clinic, Wolfson Medical Center
Other Study IDs: DD-CVD-1
Record Dates: First submitted 2007-08-05; First posted 2007-08-07 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2007-05

CONDITIONS: Infection; Acute Coronary Syndrome; Cerebrovascular Disease
Keywords: cerebro vascular event
MeSH Terms: conditions — Infections; Acute Coronary Syndrome; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The association between the levels of d-dimer, fibrinogen and PAI-1 in plasma of elderly patients admitted to internal medicine departments because of infection and the occurrence of cardio- and cerebro-vascular disease after discharge

ELIGIBILITY:
Inclusion Criteria:

* Acute infection

Exclusion Criteria:

* Anticoagulant therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients hospitalized due to infections
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
thrombosis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Asher Winder, MD, Principal Investigator — Wolfson Medical Center